CLINICAL TRIAL: NCT01399541
Title: Recovery and Rehabilitation After Lung Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Tone Rustøen, Professor, Oslo University Hospital
Other Study IDs: 59081001
Record Dates: First submitted 2010-10-01; First posted 2011-07-21 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer; Pain; Fatigue; Depression; Breathlessness
Keywords: Symptoms; Symptoms cluster; Fatigue; Depression; Sleeplessness; Social support; Stigma
MeSH Terms: conditions — Lung Neoplasms; Pain; Fatigue; Depression; Dyspnea; Sleep Initiation and Maintenance Disorders; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Under and over 65 years

SUMMARY:
The specific aims of this translational, interdisciplinary, multi-center, international research study with 300 Lung cancer patients are to:

Aim 1 Explore how the patients experience the transfer between different locations and between different levels of care at the same location and how they experienced coming home.

Aim 2 Explore lung cancer patients' symptoms, symptom clusters, and changes in symptoms and symptom clusters over time.

Aim 3 Explore interaction between lung cancers patients' symptoms, symptom clusters, health related quality of life and social support.

DETAILED DESCRIPTION:
Approximately 2500 patients are diagnosed with lung cancer annually i Norway, and approximately 400 of these undergo surgery. Many patients report that life after lung cancer surgery is difficult. After surgery, the patients are frequently transferred to a local hospital or to another level of care at the hospital where they were operated. The transfer is critical for patients' safety because communication failure is one of the most common causes of medical error.

Studies that have analyzed the quality of life of lung cancer patients after surgery reach different conclusions about the patients' Quality of life (QOL), some studies state that lung cancer patients are back to normal quality of life after 9 months, while others indicate that the patients still have reduced QOL two years after surgery. It is difficult to assess the reason for the differences in results as most of the studies used the same QOL questionnaire. Studies that have evaluated the social support that lung cancer patients receive indicate that lung cancer patients receive less support than other cancer patients.

Lung cancer patients have a wide range of physical problems (fatigue, dyspnea, coughing and pain) and psychological (depression) problems following surgery.

Based on findings from this literature review a need exist for improved postoperative follow-up of patients after surgery for lung cancer The proposed study will evaluate the social support, the levels of lung cancer stigma, symptoms and changes in this over time as well as evaluate patient experience with transfer in the immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* patients with lung cancer patients above the age of 18 that have been treated with surgery, who are able to speak and understand Norwegian,

Exclusion Criteria:

* and who suffer no cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are lung cancer patients above the age of 18 that have been treated with surgery, who are able to speak and understand Norwegian, and who suffer no cognitive impairment. The patients in the study must give written informed consent to participation in the study. It is estimated that we need 300 patients.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Key measures that will be the focus of the study is Quality of life. | 1 year with 5 measurement points
  Data will be collecetd using the self administered questionnaire: EORTC QLQ-C30 + LC13

SECONDARY OUTCOMES:
The total burden of symptoms will be one key measures in this observational study. | one year with 5 measuresments
  The self administered questionnaire: Memorial Assessment scale (MSAS) Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
A key measure to measure fatigue will be used. | one year with five measurements points
  The self administered questionnaire: Lee Fatigue Scale, LFS. Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
A key measures to measure sleep disturbances will be used. | One year with five measurements points
  A questionnaire: General sleep disturbances scale (GSDS). Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
A key measures will be used to evaluate social support | One year with two measurements points
  The self administered questionnaire: Social Provision Scale. Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
A self administered questionnaire to measure Anxiety | One year with five measurements points
  The self administered questionnaire: State and trait anxiety (STAI). Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
A self administered questionnaire to measure pain | one year with five measurements points
  The self administered questionnaire: Brief Pain Inventory. Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
Depression is a key measure | One year with five measurements points
  The self administered questionnaire: Self-report depression scale (CES-D). Key measures that will be used to evaluate the intervention(s) or, for observational studies, that are a focus of the study.
One key measures that will be used to evaluate stigma related to having lung cancer in this observational study. | 1 year with one measurements points
  Data will be collected using the self administered questionnaire: Cataldo Lung Cancer Stigma Scale (CLCSS)

CONTACTS AND LOCATIONS:
Overall Officials: Tone Rustøen, PhD, Principal Investigator — Oslo University Hospital
Locations (4):
- Norway (4):
  - Haukeland Sykehus, Bergen
  - Rikshospitalet, OUS, Oslo
  - Ullevaal University Hospital, Oslo
  - St. Olavs Hospital, Trondheim